CLINICAL TRIAL: NCT03042598
Title: Is Biphasic Ventilation Airway Management Utilizing Biphasic Cuirass Ventilation a Feasible Method to Provide Ventilation During the Apneic Phase for Patients Undergoing Emergent Rapid Sequence Intubation in the Emergency Department?
Brief Title: Biphasic Ventilation Airway Management Clinical Trial
Acronym: BVAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center of Southern Nevada (Other)
Responsible Party: Principal Investigator, David E Slattery, MD, University Medical Center of Southern Nevada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EM 2016.05
Record Dates: First submitted 2016-11-02; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Intubation
Keywords: Safe Apneic Period; Emergency Intubation; Biphasic Cuirass Ventilation (BCV); Non-invasive ventilation; Peri-intubation Hemodynamic instability; desaturation; waveform capnography; Patient safety

STUDY DESIGN:
Intervention Model Description: This is a single arm interventional feasibility trial to determine if the use of a Biphasic Cuirass Ventilator during the apneic period of intubation will decrease the prevalence of oxygen desaturation in patients undergoing RSI as compared to historical proportions of 20%.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biphasic Cuirass Ventilation (Experimental): Patients requiring emergent intubation in the Emergency Department will be provided ventilation during the apnic phase of intubation via the use of BCV.
  Interventions: Device: Biphasic Cuirass Ventilation

INTERVENTIONS:
Device: Biphasic Cuirass Ventilation — The RTX Respirator will be applied to the patient's chest to provide non-invasive ventilatory support using a Biphasic Cuirass Ventilation technology to increase the safe apnic period during intubation.
  Other Names: RTX Respirator, Hayek Medical

SUMMARY:
Investigators intend to determine if the use of Biphasic Cuirass Ventilation (BCV) improves patient safety (avoiding hypoxia) during emergency rapid sequence intubation .

DETAILED DESCRIPTION:
Methods/ Interventions:

Patients who are deemed to meet inclusion criteria and none of the exclusion criteria will be preoxygenated by any of the acceptable standard preoxygenation strategies (non-rebreather face mask, noninvasive positive pressure ventilation, etc.) . Patients will be placed and maintained on continuous 3-lead cardiac, automatic blood pressure, pulse oximeter, and waveform capnography monitoring for the duration of the procedure. Prior to induction, and during the pre oxygenation phase, subjects will be placed on the Biphasic Cuirass Ventilation (BCV) device per the manufacturer's guidelines. After adequate preoxygenation has been achieved (as determined by the treating emergency physician), the BCV assisted ventilations will be maintained and standard of care intubation procedures including apenic oxygenation if ordered by attending emergency physician will be utilized. BCV will be discontinued upon confirmation of proper tracheal intubation by waveform capnography.

Safety The BCV device covers the anterior chest wall, and therefore, it cannot be in place if CPR is needed. Therefore, all patients in cardiac arrest will be excluded. Investigators will be excluding patients with a pacemaker or central line which impairs the ability of the Curiass shell to secure on the anterior chest. Finally, patients with a history of valvular heart disease will be excluded. The protocol directs the device be applied during the normal preoxygenation period (~within that 3-5 minute period of time prior to the administration of the induction and paralytic medications). There are no other known side effects of this device. There is a potential for the device application to delay the intubation attempt; however, it is not known whether delaying intubation ,while augmenting a patient's breathing with the BCV device, negatively impacts the patient's condition. The data collection form explicitly asks the intubating physician thinks that the device delayed the intubation attempt in any way. The data collection form also tracks all of the relevant time milestones. Both of these items will be reviewed periodically during the study as safety endpoints by the data monitoring committee and will be included in the manuscript results.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the adult emergency department and require emergency intubation.
* Patient's primary language is English.

Exclusion Criteria:

* Cardiac arrest.
* Attending provider excludes patient as being at high risk for cardiac arrest or for any other reason.
* Patients who are known or reported to be pregnant pre-procedure.
* Patients in the custody of law enforcement.
* Inability to pre-oxygenate patient to an SPO2 equal to or greater than 95 percent prior to induction.
* Morbidly or Extremely obese patients defined by the NIH as BMI greater than 40.
* History of valvular heart disease.
* Presence of subclavian central line or pacemaker which impairs ability of shell to seal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-01-14 (Actual); Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Composite Primary Endpoint is the composite prevalence of any desaturation defined as SPO2 < 95% or Bradycardia, HR <60 beats per minute sustained for at least 30 seconds | 0 to 5 minutes after intubation
  The primary outcome measure is the composite prevalence of any desaturation defined as SPO2 < 95% or Bradycardia, HR <60 beats per minute sustained for at least 30 seconds, during and in the immediate post intubation (5 minutes after tracheal intubation is confirmed) period.

SECONDARY OUTCOMES:
Prevalence of post-paralytic Bag valve mask use | Time from paralytics administered until proper endotracheal tube placement is confirmed.
  Prevalence of post-paralytic administration bag valve mask ventilation in subjects enrolled into trial. We will describe this with a percentage and surrounding 95% confidence interval. This outcome reflects the potential need for ventilation during and around the intubation attempt. Our hypothesis is that BCV will eliminate the physiologic need for BVM rescue ventilation between the time paralytics are administered until the endotracheal tube is confirmed to be properly placed.
Waveform capnography pattern | Baseline to 30 minutes after intubation
  The investigators will describe the pattern of waveform capnography as measured by the research nasal capnography monitor. The waveform capnography trends will be represented graphically as continuous data for each subject over time to reflect the patterns observed from baseline until endotracheal tube is successfully placed in the trachea.
Change in End-Tidal Carbon Dioxide (ETCO2) values | Period of time from acquiring baseline ETCO2 value to successful intubation.
  We will describe the change in the mean +/- SEM and median +/- IQR ETCO2 values as measured from baseline to intubation.
Blood Pressure response to the BCV device | Baseline vital signs to 30 Minutes after intubation
  Investigators will describe the physiologic response to the BCV device by graphically representing each subject's systolic, diastolic, and mean arterial pressures (mmHG) in serial 5 minute measurements obtained from the immediate pre-application of the BCV device period until 30 minutes after intubation is complete. Unit of measure= mmHG
SpO2 response to pre-oxygenation attempts BCV application | Baseline vital signs to 30 Minutes after intubation
  Investigators will describe the physiologic response to the BCV device by graphically representing each subject's oxygen saturation measurements obtained from the immediate pre-application of the BCV device period until 30 minutes after intubation is complete. Unit of measure= % oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: David E Slattery, MD, Principal Investigator — University Medical Center of Southern Nevada
Locations (1):
- University Medical Center of Southern Nevada, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared

REFERENCES:
- [Background] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948
- [Background] Bodily JB, Webb HR, Weiss SJ, Braude DA. Incidence and Duration of Continuously Measured Oxygen Desaturation During Emergency Department Intubation. Ann Emerg Med. 2016 Mar;67(3):389-95. doi: 10.1016/j.annemergmed.2015.06.006. Epub 2015 Jul 9. PMID 26164643
- [Background] Sakles JC, Chiu S, Mosier J, Walker C, Stolz U. The importance of first pass success when performing orotracheal intubation in the emergency department. Acad Emerg Med. 2013 Jan;20(1):71-8. doi: 10.1111/acem.12055. PMID 23574475
- [Background] Brimacombe J, Keller C. Who is at increased risk of aspiration? Br J Anaesth. 2005 Feb;94(2):251; author reply 251-2. doi: 10.1093/bja/aei511. No abstract available. PMID 15629910
- [Background] Kamine TH, Papavassiliou E, Schneider BE. Effect of abdominal insufflation for laparoscopy on intracranial pressure. JAMA Surg. 2014 Apr;149(4):380-2. doi: 10.1001/jamasurg.2013.3024. PMID 24522521
- [Background] Li J, Murphy-Lavoie H, Bugas C, Martinez J, Preston C. Complications of emergency intubation with and without paralysis. Am J Emerg Med. 1999 Mar;17(2):141-3. doi: 10.1016/s0735-6757(99)90046-3. PMID 10102312
- [Background] Benumof JL, Dagg R, Benumof R. Critical hemoglobin desaturation will occur before return to an unparalyzed state following 1 mg/kg intravenous succinylcholine. Anesthesiology. 1997 Oct;87(4):979-82. doi: 10.1097/00000542-199710000-00034. No abstract available. PMID 9357902
- [Background] Corrado A, Gorini M, Melej R, Baglioni S, Mollica C, Villella G, Consigli GF, Dottorini M, Bigioni D, Toschi M, Eslami A. Iron lung versus mask ventilation in acute exacerbation of COPD: a randomised crossover study. Intensive Care Med. 2009 Apr;35(4):648-55. doi: 10.1007/s00134-008-1352-9. Epub 2008 Nov 20. PMID 19020859